CLINICAL TRIAL: NCT00324805
Title: A Phase III Randomized Trial of Adjuvant Chemotherapy With or Without Bevacizumab for Patients With Completely Resected Stage IB (≥ 4 cm) - IIIA Non-small Cell Lung Cancer (NSCLC)
Brief Title: Chemotherapy With or Without Bevacizumab in Treating Patients With Stage IB, Stage II, or Stage IIIA Non-small Cell Lung Cancer That Was Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Cancer and Leukemia Group B (Network); NCIC Clinical Trials Group (Network); North Central Cancer Treatment Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00509; NCI-2009-00509 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-0404; E1505; CDR0000475774; ECOG-E1505; E1505 (Other: ECOG-ACRIN Cancer Research Group); E1505 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Stage IB Lung Non-Small Cell Carcinoma AJCC v7; Stage IIA Lung Non-Small Cell Carcinoma AJCC v7; Stage IIB Lung Non-Small Cell Carcinoma AJCC v7; Stage IIIA Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; Gemcitabine; Pemetrexed; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (chemotherapy) (Active Comparator): Patients receive one of the following. For all, treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  REGIMEN 1: Vinorelbine ditartrate 30 mg/m2 IV on days 1 and 8, cisplatin 75 mg/m2 IV over 60 minutes on day 1 REGIMEN 2: Docetaxel 75 mg/m2 IV and cisplastin 75 mg/m2 IV on day 1 REGIMEN 3: Gemcitabine hydrochloride 1200 mg/m2 IV on days 1 and 8, cisplatin 75 mg/m2 IV on day 1 REGIMEN 4 (non-squamous histology only): Pemetrexed disodium 500mg/m2 IV and cisplatin 75 mg/m2 IV on day 1
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium; Other: Questionnaire Administration; Drug: Vinorelbine Tartrate
- Arm II (chemotherapy, bevacizumab) (Experimental): Patients receive chemotherapy as in Arm I. Patients also receive bevacizumab IV over 30-90 minutes on day 1. Treatment with bevacizumab repeats every 21 days for up to 1 year.
  Interventions: Biological: Bevacizumab; Drug: Cisplatin; Drug: Docetaxel; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Pemetrexed Disodium; Other: Questionnaire Administration; Drug: Vinorelbine Tartrate

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm II (chemotherapy, bevacizumab)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; Almita; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
Other: Questionnaire Administration — Ancillary studies
Drug: Vinorelbine Tartrate — Given IV
  Other Names: Biovelbin; Eunades; KW 2307; KW-2307; KW2307; Navelbine; Navelbine Ditartrate; NVB; Vinorelbine Ditartrate

SUMMARY:
This randomized phase III trial studies chemotherapy and bevacizumab to see how well they work compared to chemotherapy alone in treating patients with stage IB, stage II, or stage IIIA non-small cell lung cancer that was removed by surgery. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Bevacizumab also may stop the growth of non-small cell lung cancer by blocking the growth of new blood vessels necessary for tumor growth. It is not yet known whether chemotherapy is more effective with or without bevacizumab in treating non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate overall survival with chemotherapy with or without bevacizumab used in the adjuvant setting in patients with resected stage IB (>= 4 cm) - IIIA non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To evaluate disease-free survival and toxicity with chemotherapy with or without bevacizumab used in the adjuvant setting in patients with resected stage IB (>= 4 cm) - IIIA NSCLC.

CORRELATIVE OBJECTIVES:

I. To perform analyses of tissue and blood to establish factors that predict clinical outcome in patients receiving chemotherapy, with or without bevacizumab, for resected early stage NSCLC.

II. To determine whether smoking status is linked to outcome for patients with resected stage IB (>= 4 cm) - IIIA NSCLC treated with chemotherapy with or without bevacizumab in the adjuvant setting.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I (adjuvant chemotherapy without bevacizumab): Patients receive 1 of 4 chemotherapy regimens.

REGIMEN 1: Patients receive vinorelbine ditartrate intravenously (IV) over 10 minutes on days 1 and 8 and cisplatin IV over 60 minutes on day 1 immediately following vinorelbine ditartrate administration.

REGIMEN 2: Patients receive docetaxel IV over 1 hour on day 1 and cisplatin over 1 hour on day 1 immediately following docetaxel administration.

REGIMEN 3: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 and cisplatin IV over 60 minutes on day 1 immediately following gemcitabine administration.

REGIMEN 4 (non-squamous histology only): Patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 1 hour on day 1 immediately following pemetrexed disodium administration.

In all regimens, treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

ARM II (adjuvant chemotherapy with bevacizumab): Patients receive chemotherapy as in Arm I. Patients also receive bevacizumab IV over 30-90 minutes on day 1. Treatment with bevacizumab repeats every 21 days for up to 1 year.

After completion of study treatment, patients are followed up periodically for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible for this trial, patients must have undergone complete resection of their non-small cell lung cancer (NSCLC) [stage IB (>= 4 cm)] - [IIIA (T2-3N0, T1-3N1, T1-3N2] prior to enrollment; accepted types of resection will consist of lobectomy, sleeve lobectomy, bi-lobectomy or pneumonectomy; resections by segmentectomy or wedge resection will not be accepted; mediastinal lymph node sampling at specified levels is required pre-operatively (mediastinoscopy) or intraoperatively (level 7 and 4 for right sided tumors or level 7 and 5 and/or 6 for left sided tumors)
* Patients must be no less than 6 weeks (42 days) and no more than 12 weeks (84 days) post-thoracotomy at the time of randomization and must be adequately recovered from surgery
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Patients must not have received the following:

  * Prior systemic chemotherapy at any time; methotrexate (MTX) given in low doses for non-malignant conditions with last dose at least 2 weeks prior to date of registration will be allowed; other low dose chemotherapeutics for non-malignant conditions will be considered, but review by the study chair is required
  * Hormonal cancer therapy or radiation therapy as prior cancer treatment within 5 years of randomization; (prior surgery, biologic therapy, hormonal therapy, or radiation therapy for a malignancy over 5 years prior to enrollment that is now considered cured is acceptable)
* Patients must not have any history of cancer within 5 years from randomization, with the exception of in-situ carcinoma of the cervix or completely resected non-melanoma skin cancer
* Absolute neutrophil count (ANC) >= 1500 mm^3
* Platelets >= 100,000/mm^3
* Prothrombin time/international normalized ratio (INR) =< 1.5

  * Or, if patient is on therapeutic anticoagulation, prothrombin time/INR =< 3.0
* Partial thromboplastin time (PTT) =< institutional upper limit of normal (ULN) OR, if patient is on therapeutic anticoagulation, PTT must be =< 1.5 x ULN
* Total bilirubin =< 1.5 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) < 5 x upper limit of normal (ULN)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 5 x upper limit of normal (ULN)
* Serum creatinine =< 1.5 x institutional upper limit of normal (ULN)
* Urine protein should be screened by urine analysis for urine protein creatinine (UPC) ratio; for UPC ratio > 0.5, 24-hour urine protein must be obtained and the level must be < 1000 mg (1 g) for patient enrollment
* Patients with a known history of myocardial infarction or other evidence of arterial thrombotic disease (angina) will be allowed on study only if they have had no evidence of active disease for at least 12 months prior to randomization
* Patients with any history of cerebral vascular accident (CVA) or transient ischemic attack (TIA) will not be allowed on trial
* Women must not be pregnant or breast-feeding

  * All females of childbearing potential must have a blood or urine test within 2 weeks prior to randomization to rule out pregnancy
* Both fertile men and women must agree to use adequate contraceptive measures during study treatment and for at least 6 months after completion of bevacizumab
* Patients must not have any clinically significant ongoing, active or serious infection, symptomatic or uncontrolled congestive heart failure, symptomatic or uncontrolled cardiac arrhythmia or any other medical condition or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must have no history of bleeding diathesis or coagulopathy
* All patients must have a documented blood pressure (BP) with systolic =< 150 and diastolic =< 90 within 28 days of registration; patients with known hypertension must be on a stable regimen of anti-hypertensive therapy
* Patients receiving daily treatment with aspirin or non-steroidal anti-inflammatory agents (NSAIDS) are eligible; treatment with dipyridamole (Persantine), ticlopine (Ticlid), clopidogrel (Plavix) and/or cilostazol (Pletal) is not allowed; patients must have stopped taking any of these agents at least 7 days prior to randomization
* Patients must not have serious non-healing wound, ulcer, bone fracture, or have undergone a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to randomization OR core biopsy within 7 days prior to randomization
* Patients must not have a history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days prior to randomization
* Patients must not have any anticipated major surgical procedure(s) during the course of the study
* Patients must not have known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Patients may be on a stable regimen of therapeutic anticoagulation or may be receiving prophylactic anticoagulation of venous access devices, provided that coagulation studies meet entry criteria above; caution must be exercised for patients requiring anticoagulation, including treatment with low dose heparin or low molecular weight heparin for deep vein thrombosis (DVT) prophylaxis while on study
* Patients with ongoing post-operative hemoptysis (defined as bright red blood of 1/2 teaspoon or more) are not eligible; patients with pre-operative hemoptysis that has resolved post-operatively are eligible
* Patients who will receive pemetrexed (pemetrexed disodium)/cisplatin therapy must also meet the following criteria:

  * Patients assigned to pemetrexed/cisplatin therapy must NOT have squamous cell histology
  * Calculated creatinine clearance must be obtained within 2 weeks of randomization and calculated creatinine clearance (CrCl) must be >= 45 mL/min using the standard Cockcroft and Gault formula, or the measured glomerular filtration rate (GFR) using the appropriate radiolabeled method ([51]chromium-labeled ethylenediaminetetraacetic acid [51-CrEDTA] or technetium 99m diethylenetriamine-pentaacetic acid [Tc99m-DTPA]) must be used to calculate CrCl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1501 (Actual)
Dates: Start 2007-07-19 (Actual); Primary Completion 2015-10-20 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Wakelee, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1169):
- United States (1139):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Providence Hospital, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Regional Hospital, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - Saint Bernards Regional Medical Center, Jonesboro, Arkansas
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Adventist Health Cancer Care Center Chico, Chico, California
  - Community Cancer Institute, Clovis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - California Cancer Associates for Research and Excellence (cCare), Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Saint Rose Hospital, Hayward, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Northbay Cancer Center, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - University of Colorado, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - Montrose Memorial Hospital, Montrose, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Harold Leever Regional Cancer Center, Waterbury, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Lynn Regional Cancer Center - West, Boca Raton, Florida
  - Boca Raton Comprehensive Cancer Center, Boca Raton, Florida
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - Florida Hospital Memorial Medical Center, Daytona Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Florida Cancer Specialists-Gainesville Cancer Center, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - The Watson Clinic, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists-West Palm Beach, West Palm Beach, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Portneuf Medical Center, Pocatello, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - MacNeal Hospital and Cancer Center, Berwyn, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Saint Anthony Memorial Hospital, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Cottage, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - LaGrange Oncology Associates, Geneva, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Vigliotti, Antonio, P.G. M.D. (UIA Investigator), Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - DuPage Medical Group-Ogden, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Mid-Illinois Hematology Oncology Associates Limited, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Ascension Saint Vincent Anderson, Anderson, Indiana
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Premier Oncology Hematology Associates, Merrillville, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - The Community Hospital, Munster, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - MercyOne Genesis Davenport Cancer Center, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - MercyOne Waterloo Cancer Center, Waterloo, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Advent Health - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - King's Daughter's Medical Center, Ashland, Kentucky
  - Our Lady Bellefonte Hospital, Ashland, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Cancer Center of Acadiana, Lafayette, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Central Maine Medical Center, Lewiston, Maine
  - Saint Mary's Regional Medical Center, Lewiston, Maine
  - Mercy Hospital, Portland, Maine
  - Maine Center for Cancer Medicine-Scarborough, Scarborough, Maine
  - Maine General Medical Center-Thayer, Waterville, Maine
  - York Hospital, York Village, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Veterans Administration Medical Center-Baltimore, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Meritus Medical Center, Hagerstown, Maryland
  - Associates in Oncology Hematology PC -Kensington, Kensington, Maryland
  - Maryland Oncology Hematology PA-Aquilino Cancer Center, Rockville, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Beverly Hospital, Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Steward Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Commonwealth Hematology Oncology PC-Concord, Concord, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - MetroWest Medical Center-Framingham Union Hospital, Framingham, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Dana Farber Community Cancer Care-Haverhill, Haverhill, Massachusetts
  - Dana Farber-Merrimack Valley, Methuen, Massachusetts
  - Holy Family Hospital, Methuen, Massachusetts
  - Norwood Hospital, Norwood, Massachusetts
  - Berkshire Medical Center - Cancer Center, Pittsfield, Massachusetts
  - Dana Farber Community Cancer Care-Quincy, Quincy, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Dana Farber Community Cancer Care-Stoneham, Stoneham, Massachusetts
  - Noble Hospital, Westfield, Massachusetts
  - Dana Farber Community Cancer Care-Weymouth, Weymouth, Massachusetts
  - Commonwealth Hematology Oncology PC-Worcester, Worcester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Hospital, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Lapeer Regional Hospital, Lapeer, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center, Jackson, Mississippi
  - Keesler Medical Center, Keesler Air Force Base, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Veterans Administration, Columbia, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center, Jefferson City, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Institute-Summerlin Campus, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Foundation Medical Partners, Nashua, New Hampshire
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Ocean University Medical Center, Brick, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Saint Luke's Hospital-Warren Campus, Phillipsburg, New Jersey
  - Penn Medicine Princeton Health, Plainsboro, New Jersey
  - AtlantiCare Regional Medical Center -Main Campus, Pomona, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Saint Francis Medical Center, Trenton, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Memorial Medical Center-Main Campus, Las Cruces, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - New York Oncology Hematology PC - Albany, Albany, New York
  - New York Oncology Hematology PC - Albany Medical Center, Albany, New York
  - Kings County Hospital, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Veteran Affairs New York Harbor Healthcare System-Brooklyn Campus, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Coney Island Hospital, Brooklyn, New York
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - New York Oncology Hematology PC - Clifton Park, Clifton Park, New York
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Adirondack Cancer Center, Glens Falls, New York
  - Glens Falls Hospital, Glens Falls, New York
  - New York Oncology Hematology PC-Hudson, Hudson, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Garnet Health Medical Center, Middletown, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Kisco Medical Group, Mount Kisco, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Union Square, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Nyack Hospital, Nyack, New York
  - Hudson Valley Hematology Oncology Associates, Poughkeepsie, New York
  - MidHudson Regional Hospital of Westchester Medical Center, Poughkeepsie, New York
  - The Dyson Center for Cancer Care, Poughkeepsie, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Highland Hospital, Rochester, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Syracuse Veterans Administration Medical Center, Syracuse, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Oncology Hematology PC - Troy, Troy, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Veterans Administration Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Forum Health Cancer Care Center, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Mercy Physicians of Oklahoma-Lakeside, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Sky Lakes Medical Center - Cancer Treatment Center, Klamath Falls, Oregon
  - Asante Health System, Medford, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Mid-Columbia Medical Center/Celilo Cancer Center, The Dalles, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, DuBois, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - Central PA Hematology-Medical Oncology Associates PC, Lemoyne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Redeemer Health, Meadowbrook, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Chestnut Hill Health System, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Mercy Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Geisinger South Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Hematology and Oncology Associates of Rhode Island Inc, Cranston, Rhode Island
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Jones Clinic, Germantown, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Texas Health Presbyterian Hospital Dallas, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Hunter Holmes McGuire Veterans Administration Medical Center, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Pacific Cancer Research Consortium NCORP, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital-Luther Campus, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Aurora Cancer Care-Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Glendale, Glendale, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (18):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - London Regional Cancer Program, London, Ontario
  - Trillium Health Partners - Mississauga Hospital, Mississauga, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Algoma District Cancer Program Sault Area Hospital, Sault Ste. Marie, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Trillium Health Partners - Queensway Health Centre, Toronto, Ontario
  - CSSS Champlain-Charles Le Moyne, Greenfield Park, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Ireland (10):
  - Tallaght University Hospital, Dublin, Co Dublin
  - Saint Vincent's University Hospital, Dublin, Co Dublin
  - Mater Misericordiae University Hospital, Dublin, Co Dublin
  - Mater Private Hospital, Dublin, Co Dublin
  - Beaumont Hospital, Dublin, Co Dublin
  - University College Hospital Galway, Galway, Co Galway
  - Mid-Western Regional Hospital, Limerick, Co Limerick
  - University Hospital Waterford, Waterford, Co Waterford
  - Cork University Hospital, Cork
  - Saint James Hospital, Dublin
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- University Of Pretoria, Pretoria, South Africa

REFERENCES:
- [Derived] Wang Y, Sun Z, Sridhar A, Ramalingam SS, Wakelee HA, Gerber DE. Participation in lung cancer biospecimen studies: an analysis of the ECOG-ACRIN phase 3 E1505 and E5508 clinical trials. Lung Cancer. 2026 Feb 7;214:109304. doi: 10.1016/j.lungcan.2026.109304. Online ahead of print. PMID 41666849
- [Derived] Wakelee HA, Dahlberg SE, Keller SM, Tester WJ, Gandara DR, Graziano SL, Adjei AA, Leighl NB, Aisner SC, Rothman JM, Patel JD, Sborov MD, McDermott SR, Perez-Soler R, Traynor AM, Butts C, Evans T, Shafqat A, Chapman AE, Kasbari SS, Horn L, Ramalingam SS, Schiller JH; ECOG-ACRIN. Adjuvant chemotherapy with or without bevacizumab in patients with resected non-small-cell lung cancer (E1505): an open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2017 Dec;18(12):1610-1623. doi: 10.1016/S1470-2045(17)30691-5. Epub 2017 Nov 9. PMID 29129443
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between June 1, 2007 and September 20, 2013 from ECOG-ACRIN, SWOG, RTOG, CALGB, NCCTG, NCIC-CTG, NSABP, ACOSOG, and CTSU sites.
Groups:
- Arm I (Chemotherapy): Patients receive one of the following. For all, treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  REGIMEN 1: Vinorelbine ditartrate 30 mg/m2 intravenously (IV) on days 1 and 8, cisplatin 75 mg/m2 IV over 60 minutes on day 1 REGIMEN 2: Docetaxel 75 mg/m2 IV and cisplastin 75 mg/m2 IV on day 1 REGIMEN 3: Gemcitabine hydrochloride 1200 mg/m2 IV on days 1 and 8, cisplatin 75 mg/m2 IV on day 1 REGIMEN 4 (non-squamous histology only): Pemetrexed disodium 500mg/m2 IV and cisplatin 75 mg/m2 IV on day 1
  Cisplatin: Given IV
  Docetaxel: Given IV
  Gemcitabine Hydrochloride: Given IV
  Pemetrexed Disodium: Given IV
  Vinorelbine: Given IV
- Arm II (Chemotherapy, Bevacizumab): Patients receive chemotherapy as in Arm I. Patients also receive bevacizumab IV over 30-90 minutes on day 1. Treatment with bevacizumab repeats every 21 days for up to 1 year.
  Bevacizumab: Given IV
  Cisplatin: Given IV
  Docetaxel: Given IV
  Gemcitabine Hydrochloride: Given IV
  Pemetrexed Disodium: Given IV
  Vinorelbine: Given IV
Period: Overall Study
Arm/Group | Arm I (Chemotherapy) | Arm II (Chemotherapy, Bevacizumab)
Started | 749 | 752
Started Assigned Therapy | 737 | 735
Completed | 599 | 269
Not Completed | 150 | 483
Not completed — Adverse Event | 62 | 203
Not completed — Progression | 7 | 35
Not completed — Withdrawal by Subject | 51 | 174
Not completed — Death | 6 | 9
Not completed — Alternative therapy | 4 | 8
Not completed — Other complicating disease | 1 | 9
Not completed — Other reasons | 7 | 26
Not completed — Other | 0 | 2
Not completed — Did not start therapy | 12 | 17

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Arm I (Chemotherapy): Patients receive one of the following. For all, treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  REGIMEN 1: Vinorelbine ditartrate 30 mg/m2 IV on days 1 and 8, cisplatin 75 mg/m2 IV over 60 minutes on day 1 REGIMEN 2: Docetaxel 75 mg/m2 IV and cisplastin 75 mg/m2 IV on day 1 REGIMEN 3: Gemcitabine hydrochloride 1200 mg/m2 IV on days 1 and 8, cisplatin 75 mg/m2 IV on day 1 REGIMEN 4 (non-squamous histology only): Pemetrexed disodium 500mg/m2 IV and cisplatin 75 mg/m2 IV on day 1
  Cisplatin: Given IV
  Docetaxel: Given IV
  Gemcitabine Hydrochloride: Given IV
  Pemetrexed Disodium: Given IV
  Vinorelbine: Given IV
- Total: Total of all reporting groups
Arm/Group | Arm I (Chemotherapy) | Arm II (Chemotherapy, Bevacizumab) | Total
Number analyzed (Participants) | 749 | 752 | 1501
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (9.0) | 60.8 (8.7) | 60.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 374 | 381 | 755
  Male | 375 | 371 | 746
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 29 | 48
  Not Hispanic or Latino | 680 | 688 | 1368
  Unknown or Not Reported | 50 | 35 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 5 | 6
  Asian | 22 | 16 | 38
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 74 | 57 | 131
  White | 642 | 660 | 1302
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 12 | 19
Chemotherapy [Count of Participants; unit: Participants]
  Cisplatin/Vinorelbine | 187 | 190 | 377
  Cisplatin/Docetaxel | 172 | 171 | 343
  Cisplatin/Gemcitabine | 142 | 141 | 283
  Cisplatin/Pemetrexed | 248 | 249 | 497
  Unknown/Missing | 0 | 1 | 1
Histology [Count of Participants; unit: Participants]
  Squamous | 216 | 206 | 422
  Adenocarcinoma | 424 | 450 | 874
  Large cell | 22 | 16 | 38
  Bronchioloalveolar carcinoma (BAC) | 8 | 5 | 13
  Not otherwise specified (NOS) | 24 | 16 | 40
  Combined/mixed | 45 | 48 | 93
  Other | 10 | 10 | 20
  Unknown/missing | 0 | 1 | 1
Performance Status [Count of Participants; unit: Participants]
  Fully active | 439 | 440 | 879
  Ambulatory | 310 | 310 | 620
  Unknown/missing | 0 | 2 | 2
Urine protein:creatinine (UPC) ratio [Mean (Standard Deviation); unit: ratio] | 0.31 (3.10) | 0.18 (0.92) | 0.25 (2.28)
Urine protein [Mean (Standard Deviation); unit: mg/dL] | 95.26 (32.28) | 100.25 (32.28) | 97.79 (41.86)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time from randomization to death from any cause, and patients who were thought to be alive at the time of final analysis were censored at the last date of contact. The study failed to meet its primary endpoint.
Time Frame: From registration to death, up to 10 years
Population: All enrolled patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Chemotherapy) | Arm II (Chemotherapy, Bevacizumab)
Number analyzed (Participants) | 749 | 752
months | NA [NA to NA] — The median overall survival and corresponding 95% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment, i.e. a median has not been reached | 85.8 [74.9 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: Arm I (Chemotherapy) vs Arm II (Chemotherapy, Bevacizumab); Test type: Superiority; p = 0.90, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.82 to 1.19] — Arm II versus Arm I

2. Secondary Outcome: Disease-free Survival
Description: Disease-free survival (DFS) was defined as the time from randomization to an event. Events include disease recurrence, new primary of lung cancer, second primaries or death, whichever occurred first; however, it should be noted that patients with new primaries at other non-lung sites should have continued followup for recurrence of the original cancer. Patients that have not had an event reported at analysis were censored at their last date of disease assessment.
Time Frame: From registration to death, up to 10 years
Population: All enrolled patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Chemotherapy) | Arm II (Chemotherapy, Bevacizumab)
Number analyzed (Participants) | 749 | 752
months | 42.9 [36.7 to 57.0] | 40.6 [35.5 to 49.5]
Statistical Analysis 1: Comparison: Arm I (Chemotherapy) vs Arm II (Chemotherapy, Bevacizumab); Test type: Superiority; p = 0.95, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.86 to 1.15] — Arm II vs. Arm I

3. Other Pre Specified Outcome: Toxicity Rates as Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: If the difference in the rate of a particular category of toxicities between the 2 arms (N=750 per arm) is at least 5% (4% vs. 9%), 96% power can be attained assuming a significance level of 5% (two-sided Chi Square test) and that the lower toxicity rate for one arm is 4%. A difference in the rates of grade 3-5 arterial thromboembolic events and bleeding events will be monitored and assessed between the treatment arms.
Time Frame: Up to 1 year post-treatment
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Perform Analyses of Tissue and Blood to Establish Factors That Predict for Clinical Outcome in Patients Receiving Chemotherapy, With or Without Bevacizumab, for Resected Early Stage NSCLC.
Time Frame: From registration to death, up to 10 years
Population: Data for these studies were not collected
Arm/Group | Arm I (Chemotherapy) | Arm II (Chemotherapy, Bevacizumab)
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: To Determine Whether Smoking Status is Linked to Outcome for Patients With Resected Stage IB - IIIA NSCLC Treated With Chemotherapy With or Without Bevacizumab in the Adjuvant Setting.
Time Frame: From registration to death, up to 10 years
Population: Data were not collected
Arm/Group | Arm I (Chemotherapy) | Arm II (Chemotherapy, Bevacizumab)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Description: One patient who did not start treatment submitted an adverse event report
Arm/Group | Arm I (Chemotherapy) | Arm II (Chemotherapy, Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 424/738 | 563/735
Other Adverse Events (participants affected / at risk) | 474/738 | 509/735
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Chemotherapy) (N=738) | Arm II (Chemotherapy, Bevacizumab) (N=735)
Hearing impaired (Ear and labyrinth disorders) | 6 | 2
Tinnitus (Ear and labyrinth disorders) | 4 | 4
Anemia (Blood and lymphatic system disorders) | 52 | 40
Febrile neutropenia (Blood and lymphatic system disorders) | 31 | 43
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 0 | 3
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 7
Sinus tachycardia (Cardiac disorders) | 0 | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 66 | 92
Fever (General disorders) | 0 | 2
Infusion site extravasation (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 6
Pain (General disorders) | 2 | 1
Sudden death NOS (General disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 22
Cheilitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 5 | 2
Colonic hemorrhage (Gastrointestinal disorders) | 0 | 2
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 8 | 5
Diarrhea (Gastrointestinal disorders) | 15 | 31
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 2
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Esophageal pain (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 3 | 3
Mucositis oral (Gastrointestinal disorders) | 4 | 12
Nausea (Gastrointestinal disorders) | 63 | 74
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 38 | 47
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 7 | 6
Autoimmune disorder (Immune system disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1
Serum sickness (Immune system disorders) | 0 | 1
Anorectal infection (Infections and infestations) | 1 | 0
Bladder infection (Infections and infestations) | 0 | 1
Bronchial infection (Infections and infestations) | 3 | 1
Catheter related infection (Infections and infestations) | 0 | 3
Device related infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 2 | 2
Esophageal infection (Infections and infestations) | 0 | 1
Gum infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 8 | 11
Pleural infection (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 4 | 5
Skin infection (Infections and infestations) | 2 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 4 | 5
Infections and infestations - Other (Infections and infestations) | 10 | 18
Vascular access complication (Injury, poisoning and procedural complications) | 2 | 3
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 4
Alanine aminotransferase increased (Investigations) | 2 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Cardiac troponin I increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 6 | 9
INR increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 7 | 11
Neutrophil count decreased (Investigations) | 237 | 273
Platelet count decreased (Investigations) | 30 | 44
Weight loss (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 41 | 42
Investigations - Other, specify (Investigations) | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 9 | 19
Dehydration (Metabolism and nutrition disorders) | 40 | 45
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 11 | 9
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 6
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 20 | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 4
Hyponatremia (Metabolism and nutrition disorders) | 44 | 66
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 | 7
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Ataxia (Nervous system disorders) | 1 | 3
Cognitive disturbance (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 4 | 12
Dysphasia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 5 | 18
Intracranial hemorrhage (Nervous system disorders) | 1 | 1
Ischemia cerebrovascular (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 5
Reversible posterior leukoencephalopathy (Nervous system disorders) | 0 | 3
Seizure (Nervous system disorders) | 1 | 3
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 8 | 10
Nervous system disorders - Other (Nervous system disorders) | 0 | 5
Blurred vision (Eye disorders) | 1 | 1
Photophobia (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 4
Depression (Psychiatric disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory thoracic mediastinal - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 6 | 6
Chronic kidney disease (Renal and urinary disorders) | 1 | 3
Hematuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 17
Urinary retention (Renal and urinary disorders) | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 19 | 200
Hypotension (Vascular disorders) | 7 | 11
Peripheral ischemia (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 12 | 33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Chemotherapy) (N=738) | Arm II (Chemotherapy, Bevacizumab) (N=735)
Anemia (Blood and lymphatic system disorders) | 256 | 183
Fatigue (General disorders) | 62 | 68
Creatinine increased (Investigations) | 169 | 247
Neutrophil count decreased (Investigations) | 220 | 236
Platelet count decreased (Investigations) | 48 | 49
Peripheral sensory neuropathy (Nervous system disorders) | 53 | 58
Proteinuria (Renal and urinary disorders) | 3 | 48
Hypertension (Vascular disorders) | 2 | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less